CLINICAL TRIAL: NCT05590702
Title: French Observational Study of Patients With Chronic Lymphocytic Leukemia Or Small Lymphocytic Lymphoma in Real-World Settings. A FILO Study.
Brief Title: French Observational Study of Patients With Chronic Lymphocytic Leukemia Or Small Lymphocytic Lymphoma in Real-World Settings
Acronym: FOLLOW
Status: Active, not recruiting | Type: Observational
Sponsor: French Innovative Leukemia Organisation (Other)
Collaborators: AbbVie (Industry); AstraZeneca (Industry); BeiGene (Industry); Janssen-Cilag Ltd. (Industry)
Responsible Party: Sponsor
Other Study IDs: FILObsLLC_FOLLOW
Record Dates: First submitted 2022-10-17; First posted 2022-10-21 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-11

CONDITIONS: CLL/SLL

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 7 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Drug: First line therapy — Patient with CLL or SLL requiring a therapeutic strategy according to iwCLL criteria or investigator evaluation will be identified in MCM (multidisciplinary collegial meeting).
  Patients will be treated and managed according to the decision of their physicians and the related MDM. No treatment plan is recommended in the setting of this non-interventional study.

SUMMARY:
Chronic lymphocytic leukemia (CLL) is the most frequent form of leukemia in the Western World. The disease is characterized by the accumulation and proliferation of mature, monoclonal, CD5+ B-cells with specific immunophenotype in the peripheral blood (above 5x109/L), bone marrow and secondary lymphoid organs. Small lymphocytic leukemia (SLL) is characterized by similar tumor cells but without increased lymphocyte count. The management of these patients have considerably changed over the last decade. Indeed, beyond chemo-immunotherapy, multiple targeted therapies have been approved on the basis of phase 2 and randomized phase 3 clinical trials and have subsequently been used in daily practice. The management of patients with SLL is similar to that of those with CLL. In addition to therapeutic advances, the advent of new sequencing technologies has also identified CLL genetic features that are now being incorporated in patient routine evaluation.

We here propose to set a large-scale prospective and non-interventional study including patients with symptomatic CLL/SLL with the aim to evaluate the real-world clinical management of these patients and to identify the impact of treatments and therapeutic trajectories on long-term outcome.

DETAILED DESCRIPTION:
Chronic lymphocytic leukemia (CLL) is the most frequent form of leukemia in the Western World. The disease is characterized by the accumulation and proliferation of mature, monoclonal, CD5+ B-cells with specific immunophenotype in the peripheral blood (above 5x109/L), bone marrow and secondary lymphoid organs. Small lymphocytic leukemia (SLL) is characterized by similar tumor cells but without increased lymphocyte count. In Europe, CLL has been identified as the second most frequent hematological malignancies after multiple myeloma (Eurocare 5 study) and its standardized incidence in the world has been estimated to be 4/100000 person-years for men and 2.1/100000 person-years for women. In France, 4674 new cases have been observed in 2018 (FRANCIM). A proportion of patients can initially be monitored only while others with symptomatic disease at diagnosis or during follow-up require therapies. The management of these patients have considerably changed over the last decade. Indeed, beyond chemo-immunotherapy, multiple targeted therapies have been approved on the basis of phase 2 and randomized phase 3 clinical trials and have subsequently been used in daily practice. The management of patients with SLL is similar to that of those with CLL. In addition to therapeutic advances, the advent of new sequencing technologies has also identified CLL genetic features that are now being incorporated in patient routine evaluation.

Conventional chemo-immunotherapy (CIT) has been the long-standing option for CLL patient without TP53 disruption and different regimens have emerged depending on patient comorbidities (fludarabine-cyclophosphamide-rituximab, FCR; bendamustin-rituximab, BR; GA101-chloraminophene, G-CLB). These regimens fail to be effective in patients with TP53 disruption and alternative strategies are proposed for them.

The CLL therapeutic panel is now enriched by oral kinase inhibitors targeting the B-cell receptor signaling. The Bruton's tyrosine kinase inhibitors (BTKi) have been shown to provide prolonged response, even in cases where CIT usually failed, such as patients harboring TP53 disruption. In relapsed/refractory patients, median PFS with the BTKi ibrutinib is 44 months. In the frontline setting, ibrutinib has recently been shown to result in superior PFS and less infectious complications than standard CIT regimens.

The advent of the BCL2 (B-cell lymphoma 2) inhibitor venetoclax has recently added another option for the treatment of CLL patients. BCL2 is an antiapoptotic molecule governing mitochondrial apoptosis and is strongly expressed in CLL cells. Inhibiting BCL2 with venetoclax as monotherapy led to 79% response rate in the relapse/refractory setting. Combining venetoclax to rituximab demonstrated better PFS than bendamustine-rituximab in relapsed/refractory patients.

However, these treatment approaches also come with new challenges that are difficult to-address in phase 3 clinical trials and that deserve larger scale studies and longer follow-up. The emergence of drug resistance, the changes of safety profiles to deal with in routine practice and the observance of these orally administered drugs are emerging as new concerns. How these compounds change the incidence of typical CLL complication such as Richter transformation, immune cytopenias and infections remains to be determined. A growing body of concerns is also raising regarding the unlimited administration of some of this the compounds (costs, resistance, tolerance). Finally, the optimal order of use of these drugs is unknown.

The advent of the BCL2 (B-cell lymphoma 2) inhibitor venetoclax has recently added another option for the treatment of CLL patients 11,12. BCL2 is an antiapoptotic molecule governing mitochondrial apoptosis and is strongly expressed in CLL cells. Inhibiting BCL2 with venetoclax as monotherapy led to 79% response rate in the relapse/refractory setting. Combining venetoclax to rituximab demonstrated better PFS than bendamustine-rituximab in relapsed/refractory patients12.

However, these treatment approaches also come with new challenges that are difficult to-address in phase 3 clinical trials and that deserve larger scale studies and longer follow-up. The emergence of drug resistance, the changes of safety profiles to deal with in routine practice and the observance of these orally administered drugs are emerging as new concerns. How these compounds change the incidence of typical CLL complication such as Richter transformation, immune cytopenias and infections remains to be determined. A growing body of concerns is also raising regarding the unlimited administration of some of this the compounds (costs, resistance, tolerance). Finally, the optimal order of use of these drugs is unknown.

Primary objective : Setting a prospective cohort of real-world CLL/SLL patients with symptomatic disease in order to evaluate medical practices and their change and representativity over time.

Secondary objectives : Overall survival and long-term toxicity, Response and PFS at each line of therapy, Impact of therapeutic trajectories on patient outcome, Representativity of the studied population

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18-year old
* CLL or SLL requiring a therapeutic strategy according to iwCLL criteria or investigator evaluation
* Patient requiring therapy for immune events (autoimmune Thrombocytopenia and autoimmune hemolytic anemia) are eligible
* Patients who have been informed verbally and in writing about this study, and who do not object to their data being electronically processed or subjected to data quality control
* All consecutive patients for whom a discussion in the setting of local or regional multidisciplinary collegial meeting (in french : réunion de concertation pluridisciplinaire / RCP) has retained the need for starting a therapeutic strategy (curative or palliative)
* Patients with untreated or previously treated CLL/SLL are both eligible
* Patients enrolled in a clinical trial can be included in this non-interventional cohort study
* Patients requiring therapy for CLL/SLL-associated immune events only are also eligible

Exclusion Criteria:

* Patients with no need of therapy
* Patients with asymptomatic Binet A CLL
* Patient with Richter's syndrome at inclusion
* Patient requiring immunoglobulin substitution (with no need of a more specific therapy)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient with CLL or SLL requiring a therapeutic strategy according to iwCLL criteria or investigator evaluation will be identified in MCM (multidisciplinary collegial meeting).
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2022-11-11 (Actual); Primary Completion 2025-04-18 (Actual); Study Completion 2032-12-01 (Estimated)

PRIMARY OUTCOMES:
Representativity of CLL therapies and sequences across | 7-year period of time
  Number of patients who received a particular type of therapy (chemo-immunotherapy, kinase inhibitors targeting the B-cell receptor signaling, B-cell lymphoma 2 inhibitor) at baseline and in relapse and in which sequence

SECONDARY OUTCOMES:
Overall survival | 7 years
  registering cause of death focusing on CLL, infection, Richter's syndrome, immune disorders and secondary malignancies
Long-term toxicity | 7 years
  infection requiring hospitalization, secondary malignancies, cardiac and vascular events

CONTACTS AND LOCATIONS:
Overall Officials: Romain GUIEZE, Principal Investigator — French Innovative Leukemia Organisation; Xavier TROUSSARD, Study Chair — French Innovative Leukemia Organisation
Locations (57):
- France (57):
  - AMIENS - CH Amiens Picardie Site Sud, Amiens
  - Angers Chu, Angers
  - ANNECY - CH Annecy Genevois, Annecy
  - ARGENTEUIL - Centre hospitalier Victor Dupouy, Argenteuil
  - AVIGNON - Centre Hospitalier, Avignon
  - BESANCON - Hôpital Jean Minjoz, Besançon
  - BEZIERS - Centre Hospitalier - Hématologie, Béziers
  - BLOIS CH, Blois
  - APHP - Hôpital Avicenne, Bobigny
  - APHP - Hôpital Jean Verdier, Bondy
  - BOURGOUIN-JALLIEU - CH Pierre Oudot, Bourgoin
  - BREST - Hôpital Morvan - Hématologie Clinique, Brest
  - CAEN - IHBN - Hématologie Clinique, Caen
  - CERGY PONTOISE - CH René Dubos, Cergy-Pontoise
  - CHAMBERY - CH Métropole Savoie, Chambéry
  - Clermont-Ferrand - Chu Estaing, Clermont-Ferrand
  - Corbeil-Essonnes - Chsf, Corbeil-Essonnes
  - Dijon Chu, Dijon
  - GRENOBLE GHM - Institut Daniel Hollard, Grenoble
  - Grenoble - CHUGA - Hématologie Clinique, Grenoble
  - La Roche Sur Yon - Chd Vendee, La Roche-sur-Yon
  - Le Mans CH, Le Mans
  - LENS - GHT Artois, Lens
  - LIBOURNE - Hôpital Robert Boulin, Libourne
  - LILLE GHICL - Hôpital Saint Vincent de Paul, Lille
  - LILLE CHU - Hôpital Claude Huriez, Lille
  - LIMOGES - CHU Dupuytren 1, Limoges
  - LYON-Centre Léon Bérard, Lyon
  - METZ-THIONVILLE CHR- Hôpital de Mercy, Metz
  - MONTPELLIER - Hôpital Saint-Eloi - Hématologie Clinique, Montpellier
  - MORLAIX - CH des pays de Morlaix, Morlaix
  - Mulhouse - Ghrmsa, Mulhouse
  - NANTES - Hôpital Hôtel Dieu - Hématologie Clinique, Nantes
  - NIMES - CHU Caremeau, Nîmes
  - ORLEANS - CHR - Hématologie, Orléans
  - APHP - HOPITAL COCHIN - Hématologie, Paris
  - APHP - Hôpital Pitié Salpêtrière - Hématologie, Paris
  - PERPIGNAN - CH St Jean - Hématologie Clinique, Perpignan
  - Bordeaux Pessac, Pessac
  - Perigueux - Ch, Périgueux
  - LYON HCL - CH Lyon Sud, Pierre-Bénite
  - QUIMPER - CH de Cornouaille, Quimper
  - Reims Chu, Reims
  - RENNES - CHU Pontchaillou - Hématologie Clinique, Rennes
  - RENNES - Hôpital Pontchaillou - Hématologie, Rennes
  - ROUEN - Centre Henri Becquerel - Service Hématologie Clinique, Rouen
  - SAINT-BRIEUC - Hôpila Yves Le Foll, Saint-Brieuc
  - La Reunion - Gh Site Sud, Saint-Pierre
  - ST ETIENNE - CHU et Institut De Cancérologie Lucien Neuwirth, Saint-Priest-en-Jarez
  - Strasbourg - Icans, Strasbourg
  - Toulouse - IUCT Oncopole - Service d'Hématologie, Toulouse
  - TOURS - Hôpital Bretonneau, Tours
  - Troyes Ch, Troyes
  - NANCY - CHU Brabois, Vandœuvre-lès-Nancy
  - Vannes - Chba, Vannes
  - VERSAILLES - Hôpital André Mignot, Versailles
  - Villejuif Igr, Villejuif

IPD SHARING:
Plan to Share IPD: No